CLINICAL TRIAL: NCT00242372
Title: A 24-Week Randomised, Double-Blind, Multi-Centre, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Tesaglitazar Therapy When Added to the Therapy of Patients With Type 2 Diabetes Poorly Controlled on Insulin
Brief Title: GALLANT 9 Tesaglitazar vs. Placebo in Combination With Insulin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00033
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Insulin dependent Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Tesaglitazar 0.5
Drug: Insulin at least 30 units/day

SUMMARY:
This is a 24-week randomized, double-blind, multi-center, placebo-controlled study of tesaglitazar in patients with type 2 diabetes who are not adequately controlled on insulin (along or in combination with one or more oral antidiabetic agents in addition to diet and lifestyle advice). The study comprises a 3-week enrollment period and a 24-week randomized, double blind, multi-center, placebo-controlled treatment period and a 3-week follow-up. Patients must receive at least 30 units of insulin per day and will continue their current oral antidiabetic treatment regimen throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes for less than 20 years and receiving at least 30 U insulin per day

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with any thiazolidinedione class of antidiabetic agents
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2004-08; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
The change in fasting plasma glucose (FPG), insulin, proinsulin and C-peptide from baseline to the end of the randomized treatment period
Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model from baseline to the end of the randomized treatment period
Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids, lipoprotein particle size and c
C-reactive protein, LDL C/HDL C ratio and Apo B/Apo A-I ratio
FPG, homeostasis assessment model, insulin, proinsulin, C-peptide
Tumor necrosis factor-alpha, intracellular adhesion molecule-1
Fibrinogen
Urinary albumin excretion
Waist/hip ratio
Responder analyses for HbA1c, FPG, TG, HDL C, total cholesterol, non HDL C and LDL C according to pre-specified values
Proportion of patients reaching pre-specified target levels for HbA1c, FPG, TG, HDL C, non-HDL C and LDL C
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination
To validate the Work Productivity and Activity Impairment-Diabetes Questionnaire (WPAI-Diabetes) and the Diabetes Productivity Impairment Questionnaire (DPIQ) in patients with type 2 diabetes and to explore the effects of tesaglitazar (0.5 mg) on pati

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (71):
- United States (71):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tuscson, Arizona
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, La Jolla, California
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hills, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Chicago Heights, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Cadillac, Michigan
  - Research Site, Richmond Heights, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, North Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Dover, New Hampshire
  - Research Site, Roseland, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Cheswick, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Corpus Christie, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Renton, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin